CLINICAL TRIAL: NCT04980040
Title: Post Marketing Surveillance Protocol for Nesina® Tablet [Monotherapy or Combination Therapy in Type 2 Diabetic Patients]
Brief Title: A Study for Post-Marketing Surveillance of Nesina® Tablet Monotherapy or Combination Therapy in Participants With Type 2 Diabetes (T2DM) in South Korea
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Alogliptin-6001
Record Dates: First submitted 2021-07-26; First posted 2021-07-28 (Actual); Results first posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — alogliptin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nesina® Tablet: Participants with a diagnosis of Type 2 Diabetes who took Nesina® tablet (alogliptin), as prescribed by the physician, are observed in this study.
  Interventions: Drug: Alogliptin Benzoate

INTERVENTIONS:
Drug: Alogliptin Benzoate — Alogliptin benzoate tablets
  Other Names: Nesina® Tablet

SUMMARY:
The purpose of this study is to evaluate safety by determining the incidence rates of all adverse events (AEs) including serious adverse events (SAEs)/serious adverse drug reactions (ADRs), unexpected AEs and ADRs that are not reflected in the precautions for use, ADRs already known, non-serious ADRs and other safety related information among participants who have received alogliptin for type 2 diabetes mellitus.

DETAILED DESCRIPTION:
This is a long-term prospective, observational post-marketing surveillance study of alogliptin in participants with T2DM. The study assessed the safety and effectiveness of alogliptin for its approved indication within a real-world setting in South Korea.

The study will enroll approximately 3000 participants. The data is collected prospectively at the study sites and recorded in electronic case report forms (e-CRFs). All the participants are assigned to a single observational cohort:

• Nesina® Tablet

The multi-center study is conducted in South Korea. Data is collected at 13 and 26 weeks after enrollment during standard of care office visits. The overall study was conducted during re-examination period of approximately 5 years and 4 months.

ELIGIBILITY:
Inclusion Criteria:

1. Had one of the following treatments with alogliptin for the first time as an adjunct to diet and exercise to improve glycemic control:

* Monotherapy with alogliptin
* Combination therapy with the surveillance drug (alogliptin) in case of inadequate glycemic control with metformin or sulfonylurea or thiazolidinedione single therapy
* Combination therapy with the surveillance drug (alogliptin) in case of inadequate glycemic control with thiazolidinedione and metformin combination therapy
* Combination therapy with the surveillance drug (alogliptin) in case of inadequate glycemic control with insulin (single therapy or combination with metformin) therapy
* Combination therapy with metformin in patients who have no prior history of antidiabetic medication and may not achieve adequate glycemic control with monotherapy alogliptin

Exclusion Criteria:

1. Had alogliptin treatment outside of the locally approved label in Korea
2. Had a contraindication for the use of alogliptin (as described in the Korean product label)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants diagnosed with type 2 diabetes mellitus are observed.
Sampling Method: Non-Probability Sample
Enrollment: 3623 (Actual)
Dates: Start 2014-04-19 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (22):
- South Korea (22):
  - Andong
  - Anyang-si
  - Bucheon-si
  - Busan
  - Daegu
  - Daejeon
  - Gimhae
  - Gongju
  - Goyang-si
  - Gwangju
  - Gyeongju
  - Incheon
  - Jeonju
  - Namyangju
  - Osan
  - Seongnam
  - Seongnam-si
  - Seoul
  - Suncheon
  - Suwon
  - Ulsan
  - Wŏnju

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 81 investigative sites in South Korea during the re-examination period: 19 April 2014 to 30 August 2019.
Pre-assignment Details: This post-marketing surveillance (PMS) study was conducted during a re-examination period of approximately 5 years and 4 months to investigate the safety and efficacy of monotherapy or combination therapy with alogliptin in participants with type 2 diabetes in routine care settings.
Groups:
- Nesina® Tablet: Participants with a diagnosis of Type 2 Diabetes who took Nesina® tablet (alogliptin), as prescribed by the physician, were observed in this study.
Period: Overall Study
Arm/Group | Nesina® Tablet
Started | 3623
Completed | 3131
Not Completed | 492
Not completed — Violated the Inclusion Criteria | 260
Not completed — Violated the Administration & Dosage | 225
Not completed — Lost to Safety-Follow-up | 4
Not completed — Administered the study drug prior to signing the informed consent form | 3

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included participants who were treated with the surveillance drug at least once and completed the follow-up for safety.
Arm/Group | Nesina® Tablet
Number analyzed (Participants) | 3131
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.07 (12.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1322
  Male | 1809
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3131
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Korea, Republic Of | 3131

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: An SAE is an adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. 95% Confidence Interval was calculated using exact method.
Time Frame: From first dose of study drug up to 30 days post last dose of study drug (Up to 79.77 weeks)
Population: Safety Set included all participants who had been administered the study drug and completed the follow-up.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nesina® Tablet
Number analyzed (Participants) | 3131
percentage of participants | 1.18 [0.83 to 1.63]

2. Primary Outcome: Percentage of Participants With Serious Adverse Drug Reactions (ADRs)
Description: Serious ADRs are defined as SAEs that are, in the investigator's opinion, of causal relationship to the study treatment. An SAE is an adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. 95% Confidence Interval was calculated using exact method.
Time Frame: From first dose of study drug up to 30 days post last dose of study drug (Up to 79.77 weeks)
Population: Safety Set included all participants who had been administered the study drug and completed the follow-up.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nesina® Tablet
Number analyzed (Participants) | 3131
percentage of participants | 0.16 [0.05 to 0.37]

3. Primary Outcome: Percentage of Participants With Unexpected Adverse Events
Description: An unexpected AE is an AE with a difference in nature, severity, specificity, or outcome, compared to the product licensure/safety notification of the drug. 95% Confidence Interval was calculated using exact method.
Time Frame: From first dose of study drug up to 30 days post last dose of study drug (Up to 79.77 weeks)
Population: Safety Set included all participants who had been administered the study drug and completed the follow-up.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nesina® Tablet
Number analyzed (Participants) | 3131
percentage of participants | 8.88 [7.91 to 9.93]

4. Primary Outcome: Percentage of Participants With Unexpected Adverse Drug Reactions (ADRs)
Description: Unexpected ADRs are unexpected AEs that are, in the investigator's opinion, of causal relationship to the study treatment. 95% Confidence Interval was calculated using exact method.
Time Frame: From first dose of study drug up to 30 days post last dose of study drug (Up to 79.77 weeks)
Population: Safety Set included all participants who had been administered the study drug and completed the follow-up.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nesina® Tablet
Number analyzed (Participants) | 3131
percentage of participants | 2.01 [1.55 to 2.57]

5. Secondary Outcome: Haemoglobin (HbA1c) Levels
Description: HbA1c are glycated haemoglobin or amount of glucose attached to haemoglobin.
Time Frame: Baseline (Before administration of alogliptin), 13 weeks (±2 weeks) and 26 weeks (±2 weeks) after administration
Population: Participants from the Efficacy Set, included participants who completed study drug treatment for a period exceeding 13 weeks, at the investigator's clinical judgment, with data available for analyses. Number analyzed are participants with data available for analyses at the given timepoint.
Measure: Mean (Standard Deviation); unit: percentage of Hb1Ac
Arm/Group | Nesina® Tablet
Number analyzed (Participants) | 1738
percentage of Hb1Ac
  Before Administration | 8.05 (1.48)
  13 weeks (±2 weeks) After Administration: number analyzed (Participants) | 1099
  13 weeks (±2 weeks) After Administration | 6.96 (1.08)
  26 weeks (±2 weeks) After Administration: number analyzed (Participants) | 871
  26 weeks (±2 weeks) After Administration | 6.87 (0.97)

6. Secondary Outcome: Fasting Blood Glucose Levels
Time Frame: Baseline (Before administration of alogliptin), 13 weeks (±2 weeks) and 26 weeks (±2 weeks) after administration
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Nesina® Tablet
Number analyzed (Participants) | 1681
g/dL
  Before Administration | 166.22 (58.14)
  13 weeks (±2 weeks) After Administration: number analyzed (Participants) | 1085
  13 weeks (±2 weeks) After Administration | 136.84 (38.78)
  26 weeks (±2 weeks) After Administration: number analyzed (Participants) | 871
  26 weeks (±2 weeks) After Administration | 133.09 (34.73)

7. Secondary Outcome: Percentage of Participants With HbA1c < 7.00%
Description: HbA1c are glycated haemoglobin or amount of glucose attached to haemoglobin.
Time Frame: Baseline (Before administration of alogliptin), 13 weeks (±2 weeks) and 26 weeks (±2 weeks) after administration
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Nesina® Tablet
Number analyzed (Participants) | 1738
percentage of participants
  Before Administration | 17.84
  13 weeks After Administration: number analyzed (Participants) | 1099
  13 weeks After Administration | 60.96
  26 weeks After Administration: number analyzed (Participants) | 871
  26 weeks After Administration | 63.49

8. Secondary Outcome: Percentage of Participants With Overall Improvement and Final Effectiveness Assessment
Description: Participants were assessed for overall improvement and effectiveness assessments as per the following categories: 'Improved - signs and symptoms are significantly improved'; 'Unchanged - improvement in signs and symptoms is not significant or there is no change in signs and symptoms'.
Time Frame: Up to Week 26
Population: Efficacy Set included participants who completed study drug treatment for a period exceeding 13 weeks, at the investigator's clinical judgment.
Measure: Number; unit: percentage of participants
Arm/Group | Nesina® Tablet
Number analyzed (Participants) | 1784
percentage of participants
  Improved | 82.57
  Unchanged | 9.64
  Worsened | 7.79

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days post last dose of study drug (Up to 79.77 weeks)
Description: Safety Set included all participants who had been administered the study drug and completed the follow-up.
Arm/Group | Nesina® Tablet
All-Cause Mortality (participants affected / at risk) | 0/3131
Serious Adverse Events (participants affected / at risk) | 37/3131
Other Adverse Events (participants affected / at risk) | 0/3131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nesina® Tablet (N=3131)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1
Fracture (Musculoskeletal and connective tissue disorders) | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1
Fracture lower limb (Musculoskeletal and connective tissue disorders) | 1
Fracture upper limb (Musculoskeletal and connective tissue disorders) | 1
Fracture vertebral (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis aggravated (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhagic (Gastrointestinal disorders) | 1
Appendicitis (Gastrointestinal disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Diabetes mellitus aggravated (Metabolism and nutrition disorders) | 2
Acidosis (Metabolism and nutrition disorders) | 1
Abscess (Infections and infestations) | 2
Infection (Infections and infestations) | 1
Wound dehiscence (Infections and infestations) | 1
Pulmonary carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Thyroid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pulmonary carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Back ache (General disorders) | 1
Oedema generalised (General disorders) | 1
Weakness generalized (General disorders) | 1
Asthma aggravated (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aggravated (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Kidney stone (Renal and urinary disorders) | 1
Renal function abnormal (Renal and urinary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Anorexia (Psychiatric disorders) | 2
Cerebral infarction (Vascular disorders) | 1
Transient ischaemic attack (Vascular disorders) | 1
Fibrillation atrial aggravated (Cardiac disorders) | 1
Laceration (Infections and infestations) | 1
Dysarthria (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/40/NCT04980040/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT04980040/SAP_001.pdf